CLINICAL TRIAL: NCT04994990
Title: Effective OnabotulinumtoxinA Dose Response Study for Upper Facial Wrinkles
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: staff not available to support study
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 23-0015-NH
Record Dates: First submitted 2021-08-03; First posted 2021-08-06 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Rhytides
Keywords: Botox; Facial Wrinkles; OnabotulinumtoxinA; Cosmetic; Dosage
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Dosing Group (Active Comparator)
  Interventions: Drug: OnabotulinumtoxinA Standard Dose
- Half Standard Dosing Group (Experimental)
  Interventions: Drug: OnabotulinumtoxinA Half Standard Dose

INTERVENTIONS:
Drug: OnabotulinumtoxinA Standard Dose — Active comparator group will be treated for full upper face wrinkles with standard recommended doing of onabotulinumtoxinA
  Arms: Standard Dosing Group
Drug: OnabotulinumtoxinA Half Standard Dose — Experimental group will be treated for full upper face wrinkles with half of the standard recommended doing of onabotulinumtoxinA
  Arms: Half Standard Dosing Group

SUMMARY:
This research is being done to determine if lower doses of botox than what is currently recommended can give similar results to patients, at lower cost and lower risk to them. Subjects will receive botox in the same areas of the upper face with standard doses on one side of the face. On the other side, double the botox concentration will be administered, free of charge to the participant, in order to see if the difference in concentration creates a difference in wrinkle reduction and participant satisfaction over time.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18-65
* In good general health as evidenced by medical history and exhibiting upper facial wrinkles on physical examination
* Agreement to adhere to Lifestyle Considerations (see section 5.3) as appropriate throughout study duration

Exclusion Criteria:

* Current use of aminoglycosides, curare like agents, and muscle relaxants
* Pregnancy or lactation
* Known allergic reactions to components of the botox formulation and any of its ingredients
* Treatment with another botox product for the face within 4 months
* Infections/preexisting weakness at the proposed injection sites on physical examination
* History of neuromuscular disorder, pre existing severe cardiovascular disease, compromised respiratory function, severe dysphagia
* Pediatric population, patients older than 65 since the effect of botox in terms of duration and magnitude is highly variable in these age groups.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Upper Face Wrinkle Severity 1 Week After Botox Administration | 4 Months
  The severity of upper face wrinkles will be assessed on a 0 - 4 scale by a trained observer in both relaxed and expressive states. Efficacy will be assessed at 1 week, 1 month, 2 months, 3 months, and 4 months.
Upper Face Wrinkle Severity 1 Month After Botox Administration | 4 Months
  The severity of upper face wrinkles will be assessed on a 0 - 4 scale by a trained observer in both relaxed and expressive states. Efficacy will be assessed at 1 week, 1 month, 2 months, 3 months, and 4 months.
Upper Face Wrinkle Severity 2 Months After Botox Administration | 4 Months
  The severity of upper face wrinkles will be assessed on a 0 - 4 scale by a trained observer in both relaxed and expressive states. Efficacy will be assessed at 1 week, 1 month, 2 months, 3 months, and 4 months.
Upper Face Wrinkle Severity 3 Months After Botox Administration | 4 Months
  The severity of upper face wrinkles will be assessed on a 0 - 4 scale by a trained observer in both relaxed and expressive states. Efficacy will be assessed at 1 week, 1 month, 2 months, 3 months, and 4 months.
Upper Face Wrinkle Severity 4 Months After Botox Administration | 4 Months
  The severity of upper face wrinkles will be assessed on a 0 - 4 scale by a trained observer in both relaxed and expressive states. Efficacy will be assessed at 1 week, 1 month, 2 months, 3 months, and 4 months.
Patient Satisfaction 1 Week After Botox Administration | 4 Months
  A satisfaction survey (on a scale of 0-10) will be administered to the participant at 1 week, 1 month, 2 months, 3 months and 4 months from the date of botox administration
Patient Satisfaction 1 Month After Botox Administration | 4 Months
  A satisfaction survey (on a scale of 0-10) will be administered to the participant at 1 week, 1 month, 2 months, 3 months and 4 months from the date of botox administration
Patient Satisfaction 2 Months After Botox Administration | 4 Months
  A satisfaction survey (on a scale of 0-10) will be administered to the participant at 1 week, 1 month, 2 months, 3 months and 4 months from the date of botox administration
Patient Satisfaction 3 Months After Botox Administration | 4 Months
  A satisfaction survey (on a scale of 0-10) will be administered to the participant at 1 week, 1 month, 2 months, 3 months and 4 months from the date of botox administration
Patient Satisfaction 4 Months After Botox Administration | 4 Months
  A satisfaction survey (on a scale of 0-10) will be administered to the participant at 1 week, 1 month, 2 months, 3 months and 4 months from the date of botox administration

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Bastidas, MD, Principal Investigator — Northwell Health

IPD SHARING:
Plan to Share IPD: No